CLINICAL TRIAL: NCT07330505
Title: Transducer Levelling Errors in Everyday ICU Practice - A Multicentre Blinded Observational Study
Status: Not yet recruiting | Type: Observational
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Principal Investigator, Carl Sjödin, Principal Investigator, Vastra Gotaland Region
Other Study IDs: 2024-06578-01
Record Dates: First submitted 2025-12-18; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Critically Ill; Haemodynamic Instability
Keywords: Invasive arterial blood pressure monitoring; Central venous pressure monitoring; Pressure transducer leveling; Pressure transducer positioning; Intensive care unit; Critically ill; Patient safety; Mean arterial pressure; Right atrial pressure
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Invasive Pressure Monitoring Cohort: Mechanically ventilated adult ICU patients undergoing routine invasive arterial blood pressure and central venous pressure monitoring. Pressure transducer positioning and associated pressure deviations are observed using blinded reference sensors without altering clinical care.

SUMMARY:
Invasive pressure monitoring (arterial blood pressure via arterial catheter and central venous pressure via central venous catheter) is fundamental to clinical decision-making in intensive care. Treatment with vasopressors, fluids, and nursing interventions depends on accurate measurements. Because pressure transducers are hydrostatic, even small levelling errors can produce clinically relevant deviations (approximately 1 mmHg per 1.3 cm of vertical misplacement). Such errors may contribute to inappropriate therapy, for example under-recognition of hypotension, unnecessary vasopressor escalation, or missed venous congestion.

This prospective, multicenter, blinded observational study will quantify transducer levelling deviations during routine ICU care and evaluate whether clinically relevant deviations are associated with treatment decisions. Adult mechanically ventilated ICU patients with an arterial catheter, a central venous catheter, and ongoing vasopressor therapy will be included at hospitals in Västra Götalandsregionen, Sweden. Two blinded reference lines/sensors will be placed at predefined physiological zero levels for MAP and CVP and connected in parallel to the patient monitoring system. Continuous deviation (mmHg) between the clinical transducer position and the blinded reference level will be recorded for 8 hours while clinical staff remain unaware of the reference setup. MAP/CVP-related treatment decisions (e.g., vasopressor adjustments, fluid therapy, and nursing interventions) will be recorded with timestamps.

The study will provide real-world data on the magnitude and frequency of invasive pressure transducer misalignment in daily ICU practice and its potential relationship to patient management.

DETAILED DESCRIPTION:
This is a prospective, multicenter, blinded observational study evaluating the accuracy of invasive pressure transducer levelling for arterial pressure (mean arterial pressure, MAP) and central venous pressure (CVP) during routine intensive care. Adult mechanically ventilated ICU patients with an indwelling arterial catheter and central venous catheter receiving vasopressor therapy are observed without any protocol-mandated changes to standard clinical care.

To quantify levelling deviations without influencing clinical behavior, a parallel reference measurement setup is connected to the existing monitoring system. Two fluid-filled reference lines are connected in parallel to the pressure dome used for invasive monitoring and secured to the chest wall at the fourth intercostal space at half of the anteroposterior thoracic diameter, one on each side of the chest. This configuration allows continuous estimation of vertical deviation (mmHg) between the clinical transducer position and a predefined physiological reference level. During lateral positioning, deviation is calculated using the midpoint between the two reference lines as the reference. Reference lines are covered with dressings to maintain blinding of clinical staff to the reference levels.

Physiological waveforms and calculated deviations are recorded continuously for an 8-hour monitoring period for each participant. In parallel, treatment actions plausibly influenced by interpretation of MAP or CVP (including vasopressor titration, fluid administration or removal, and nursing interventions related to positioning or transducer handling) are documented with timestamps to allow temporal association analyses. Relevant contextual variables are collected to support interpretation of deviations and clinical responses.

Data quality is ensured through predefined measurement procedures, continuous digital waveform acquisition, synchronization of reference and clinical signals, and post hoc review of signal integrity. Periods affected by technical artifacts or signal loss are flagged according to predefined criteria. Data segments that are missing, uninterpretable, or invalid due to technical failure are treated as missing and excluded from analyses, without imputation.

The study is designed to quantify the magnitude and frequency of invasive pressure transducer misalignment during routine ICU care and to explore whether clinically relevant deviations are associated with contemporaneous treatment decisions, with the aim of informing patient safety and quality improvement initiatives.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* ICU admission
* Mechanically ventilated
* Arterial catheter for MAP
* Central venous catheter for CVP
* Ongoing vasopressor therapy

Exclusion Criteria:

* Severe hemodynamic or respiratory instability
* Contraindications for lateral positioning
* Expected survival <24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult (≥18 years) critically ill, mechanically ventilated ICU patients receiving routine invasive arterial blood pressure and central venous pressure monitoring, often under sedation and vasoactive support.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Mean deviation in transducer position for MAP and CVP | During the 8-hour continuous monitoring period following initiation of blinded reference monitoring
  Continuous deviation (mmHg) between the clinical transducer position and the blinded reference zero point. Continuous (mmHg).

SECONDARY OUTCOMES:
Frequency of clinically relevant deviations | During the same 8-hour continuous monitoring period following initiation of blinded reference monitoring
  Proportion of monitoring time (%) with deviation >2 mmHg (CVP) or >5 mmHg (MAP). Percentage of total monitoring time.
Association between deviations and treatment decisions | During the 8-hour continuous monitoring period, with treatment decisions assessed within 5 minutes following detection of a deviation
  Relationship between deviation size and treatment decisions (vasopressor adjustments, fluid therapy, nursing interventions). Binary outcome (decision yes/no), regression analysis.
Differences in deviation magnitude and frequency across hospitals and ICU specialties. | During the 8-hour continuous monitoring period following initiation of blinded reference monitoring
  Differences in deviation magnitude and frequency across hospitals and ICU specialties. Continuous (mmHg), categorical (% above threshold).
Hemodynamic context of deviations | At baseline and during the subsequent 8-hour continuous monitoring period
  Association between deviation magnitude and concurrent patient status (SOFA, MAP, CVP, CO, SVR, temperature). Continuous and categorical variables.

CONTACTS AND LOCATIONS:
Overall Officials: Lotta Johansson, PhD, Principal Investigator — Sahlgrenska University Hospital

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data underlying the results will be shared on reasonable request. Shared data will be limited to variables necessary to reproduce the primary analyses and will not include any direct identifiers.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: SD: 2028-01-01 ED: 2033-12-31
Access Criteria: Access to de-identified individual participant data will be provided to qualified researchers upon reasonable request. Requests must include a brief research proposal and a data management plan. Data will be shared under a data use agreement that prohibits re-identification of participants and limits use to the approved purpose.

REFERENCES:
- [Background] 1. Cecconi, M., et al., Consensus on circulatory shock and hemodynamic monitoring. Task force of the European Society of Intensive Care Medicine. Intensive Care Med, 2014. 40(12): p. 1795-815. 2. Vincent, J.L., Critical care - where have we been and where are we going? New England Journal of Medicine, 2013. 369(19): p. 1839-1841. 3. Vincent, J.L. and D. De Backer, Circulatory shock. New England Journal of Medicine, 2013. 369(18): p. 1726-1734. 4. Giusti, G.D., Critical care nurses' perspectives on cardiac monitoring: barriers and training needs. BMC Nursing, 2024. 23: p. 742. 5. Alastalo, T.T., Critical care nurses' observational skills in detecting early patient deterioration. Intensive and Critical Care Nursing, 2017. 43: p. 97-103. 6. Magder, S., Right Atrial Pressure in the Critically Ill: How to Measure, What Is the Value, What Are the Limitations? Chest, 2017. 151(4): p. 908-916. 7. Sjödin, C., S. Sondergaard, and L. Johansson, Variability in alignment of central venous pressure transducer to physiologic reference point in the intensive care unit-A descriptive and correlational study. Aust Crit Care, 2019. 32(3): p. 213-217. 8. Figg, K.K. and E.C. Nemergut, Error in central venous pressure measurement. Anesth Analg, 2009. 108(4): p. 1209-11. 9. Oh, C., et al., Errors in pressure measurements due to changes in pressure transducer levels during adult cardiac surgery: a prospective observational study. BMC Anesthesiol, 2023. 23(1): p. 8. 10. Jacobs, K., et al., Accuracy of intra-arterial line transducer levelling practice in a general intensive care unit. Aust Crit Care, 2024. 37(1): p. 51-57.